CLINICAL TRIAL: NCT01787370
Title: Mainz Registry of Flow-mediated Constriction
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Prof., Johannes Gutenberg University Mainz
Other Study IDs: Flow-MEC
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease, endothelial dysfunction
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing coronary angiography: Consecutive patients referred for coronary angiography for the suspect of coronary artery disease

SUMMARY:
The goal of the flow-mediated constriction/ FMC-registry is to investigate whether the measurement of endothelial function using flow-mediated dilation and flow-mediated constriction provides on the presence of coronary atherosclerosis and on the prognosis of patients undergoing coronary angiography.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a lifelong process resulting from the interaction of many risk factors, environmental influences, and genetic predisposition. Although the collection of medical history and standard risk factors provides essential information, the existence of complex interactions among different risk factors, risk modifications by medical therapy, and inter-individual differences complicate these issues. In the light of these limitations, alternative approaches have been sought, and the non-invasive assessment of endothelial function has been proposed as a possible non-invasive and inexpensive endpoint that could reflect the cumulative cardiovascular burden and/or the responsiveness to therapies at the level of individual patients.

A total of 1000 consecutive patients undergoing elective coronary angiography will be studied. Patients have chest pain on effort according to the American College of Cardiology/American Heart Association 2007 Guidelines and/or a pathological exercise or dobutamine stress test. Patients undergoing catheterization for any reason other than stable (suspected) CAD (e.g. for hypertensive crisis associated with troponin elevation, or acute coronary syndromes, valvular heart disease, congenital heart disease, cardiomyopathy, etc.) will be excluded. Patients with known chronic inflammatory diseases, dialysis, or decompensated/severe heart failure will be also excluded.

Blood samples will be drawn from all patients after a fasting period of at least 12 h and will be examined with the use of routine laboratory methods for blood counts, lipid parameters, C-reactive protein, renal and hepatic function. Coronary risk factors were defined as: obesity (body mass index >30 kg/m2); age; smoking (or previous smoking); hyperlipidaemia (total serum cholesterol >220 mg/dL and/or serum triglycerides >200 mg/dL); hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg on two consecutive seated measurements or therapy with antihypertensive medication); family history (first-degree relatives with cardiovascular disease); diabetes mellitus (fasting serum glucose levels >126 mg/dL or therapy with oral hypoglycaemic agents or insulin).

The methods employed for L-FMC/FMD (flow mediated dilation)'analysis in our laboratory have been previously published (Gori Journal of the American College of Cardiology 2008). Briefly, patients will be placed supine, the left arm immobilized, and L-FMC and FMD will be measured using a Vivid 7 (General Electrics, Munich, Germany) ultrasound platform equipped with a 14 MHz matrix probe and a micrometric probe holder. Low-flow-mediated constriction corresponds to the constriction observed during a 4.5 min occlusion of a pneumatic cuff placed distal to the site of arterial diameter measurement. Flow-mediated dilation corresponds to the maximal dilation observed in the 5 min following deflation of the cuff, i.e. during reactive hyperaemia. Repeatability and reproducibility data of these methods have been recently reported (intra-class correlation coefficient=0.68 and 0.80 for FMD and L-FMC, respectively).

All data will be acquired digitally and analysed in a randomized, blinded fashion prior to coronary angiography by an investigator not aware of the clinical status of the patient, using automatic dedicated software.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* capacity to provide informed consent

Exclusion Criteria:

* Patients undergoing catheterization for any reason other than stable (suspected) CAD (e.g. for hypertensive crisis associated with troponin elevation, or acute coronary syndromes, valvular heart disease, congenital heart disease, cardiomyopathy, etc.).
* Patients with known chronic inflammatory diseases, dialysis, or decompensated/severe heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing coronary angiography for the suspect of coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2009-09; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Baseline
  Flow-mediated constriction (change in diameter of the radial artery induced by a reduction in local shear stress) will be measured at entry in the registry

SECONDARY OUTCOMES:
Endothelial function | Baseline
  Flow-mediated dilation (change in diameter of the radial artery in response to increases in shear stress) will be measured at entry in the registry

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Gori, MD PhD, Principal Investigator — Universitätsmedizin Mainz
Locations (1):
- University Medical Center Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Result] Gori T, Muxel S, Damaske A, Radmacher MC, Fasola F, Schaefer S, Schulz A, Jabs A, Parker JD, Munzel T. Endothelial function assessment: flow-mediated dilation and constriction provide different and complementary information on the presence of coronary artery disease. Eur Heart J. 2012 Feb;33(3):363-71. doi: 10.1093/eurheartj/ehr361. Epub 2011 Sep 14. PMID 21920964